CLINICAL TRIAL: NCT05554224
Title: Integrated Multi-omics and Machine Learning-driven Personalized Treatment of Obesity-associated Fatty Liver Disease
Brief Title: Integrated Multi-omics Data for Personalized Treatment of Obesity-associated Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Hospital Universitari Sant Joan (Unknown); La Caixa Foundation (Other); Instituto de Salud Carlos III (Other Government); University of Barcelona (Other)
Responsible Party: Principal Investigator, Jorge Joven, Professor of Medicine at the Rovira i Virgili University, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: EOM study; EPIMET (Other: Hospital Universitari Sant Joan)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: NAFLD; Obesity, Morbid; Comorbidities and Coexisting Conditions
Keywords: Weight loss; Bariatric surgery; Liver diseases; Mass spectrometry; Proteomics; Lipidomics; Metabolomics; Transcriptomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid; Weight Loss; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, hepatic, subcutaneous and visceral adipose tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Severe obesity without liver disease: Patients with severe obesity who did not meet the criteria described in Kleiner et al. (2005) for nonalcoholic steatohepatitis diagnosis (score 0-2).
  Interventions: Diagnostic Test: To propose diagnostic tests for liver diseases before surgical decisions.
- Severe obesity with liver disease without criteria for steatohepatitis: Patients with severe obesity who did not meet the criteria described in Kleiner et al. (2005) for nonalcoholic steatohepatitis diagnosis, but their biopsies presented some liver severity (scores 3 and 4).
  Interventions: Diagnostic Test: To propose diagnostic tests for liver diseases before surgical decisions.
- Severe obesity with well-defined steatohepatitis and/or cirrhosis: Patients with severe obesity who met the criteria described in Kleiner et al. (2005) for nonalcoholic steatohepatitis diagnosis (score 5-8).
  Interventions: Diagnostic Test: To propose diagnostic tests for liver diseases before surgical decisions.

INTERVENTIONS:
Diagnostic Test: To propose diagnostic tests for liver diseases before surgical decisions. — Observational although patients are candidates for metabolic surgery.
  Other Names: External follow up monitoring liver diseases and weight loss.

SUMMARY:
The investigators seek to analyze the samples provided by patients with obesity-associated fatty liver disease at the multi-omics level and to integrate the results with clinical information, genotypic variants, and factors influencing inter-organ crosstalk. The main aim is to improve the interpretation of fatty liver disease associated with obesity and diabetes by developing predictive models built with algorithms from artificial intelligence. The challenge is to decipher the flow of information by exploring contributing factors, proximate causes of regulatory defects, and maladaptive responses that may promote therapeutic approaches.

DETAILED DESCRIPTION:
The investigators study the most prevalent liver disease in the history of humankind, which is the leading cause of liver transplantation in its severe forms. It results from two silent pandemics with enormous health impacts: obesity and diabetes. Together or separately, they affect more than 30% of the world's population. The current term for the disease is MAFLD (metabolic (dysfunction)-associated fatty liver disease). This designation indicates that metabolic disorders related to obesity, diabetes, dyslipidemia, and hypertension are its primary cause. These disorders are related and lead to fat accumulation in the liver, the first step in a broad spectrum of chronic liver diseases. These diseases respond clinically in a very variable way and remain undiagnosed and untreated for a long time. There is no accepted pharmacological treatment, and lifestyle changes, although possibly effective, usually fail because they require particularly favorable conditions. Therefore, the identified problems that should be solve are:

(1) The diagnosis of MAFLD requires a liver biopsy, a costly and aggressive procedure. (2) Without examining the liver, clinicians can know little about the progression of the disease and the underlying causes. (3) The results in experimental models can be informative but difficult to translate to the clinic. Recent reports suggest the essential role of phospholipid biosynthesis and transport between the endoplasmic reticulum and mitochondria. (4) All of the above makes it difficult to obtain the necessary information to propose changes in clinical guidelines.

Considering these aspects, patients with morbid obesity can be an informative human model. Among other advantages, patients have surgical options that allow us to obtain portions of affected organs that facilitate specific diagnosis and that, because they require constant care, can be studied on an ongoing basis. The presented approach can improve patient care and essentially consists of identifying the most significant number of variables that can help. In particular, here are proposed the inclusion of variables that can already be obtained from recent advances in the laboratory, encompassed within the omics sciences (genomics, transcriptomics, proteomics, metabolomics, lipidomics, microbiomics). Each of these has its advantages and limitations. Predictive models can integrate these variables into clinical data to explore organ crosstalk.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater or equal to 40 kg/m^2.
* Body mass index between 35 and 40 kg/m^2 with high-risk comorbidities (diagnosis or treatment for hypertension, dyslipidemia, or type 2 diabetes mellitus).
* Positive psychiatric evaluation.
* Age greater or equal to 18 years old.

Exclusion Criteria:

* Legal or illegal drug consumption, including alcohol.
* Diagnosis of Hepatitis.
* Current cancer diagnosis or treatment.
* Clinical or analytical evidence of severe illness.
* Clinical or analytical evidence of chronic or acute inflammation.
* Clinical or analytical evidence of infectious diseases.
* Clinical or analytical evidence of terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are consecutive patients with obesity type II or III attending the bariatric surgery unit for treatment. In this center, women are more frequent than men. The average age is 49 (interquartile range 41 - 58). Steatohepatitis (~30 percent), type 2 diabetes mellitus (~40 percent), hypertension (~60 percent), and dyslipidemia (~35 percent) are the most prevalent comorbidities. Other common ailments are obstructive sleep apnea (~20 percent) and hypothyroidism (~10 percent).
Sampling Method: Probability Sample
Enrollment: 1104 (Estimated)
Dates: Start 2008-06-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | 1 to 10 years
  The effect of bariatric surgery on adiposity outcomes.
Type 2 diabetes mellitus incidence | 1 to 10 years
  The effect of bariatric surgery on metabolic outcomes.
Hypertension incidence | 1 to 10 years
  The effect of bariatric surgery on metabolic outcomes.
Chronic liver diseases incidence | 1 to 10 years
  The usefulness of imaging techniques on metabolic outcomes.
Dyslipidemia incidence | 1 to 10 years
  The effect of bariatric surgery on metabolic outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Joven, Professor, Principal Investigator — Institut Investigacio Sanitaria Pere Virgili
Locations (1):
- Hospital Universitari Sant Joan, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The Data Management Plan makes data fully findable, accessible, interoperable, and reusable, following the indication of the Horizon 2020 initiative of the European Union. The clinical team identified sensitive data, including epidemiological, anthropometric, and medical information. It is the only responsibility of the principal investigator to ensure that sensitive data are de-identified, implementing technical safeguards to guarantee anonymity.
  Most data will be experimental and obtained from the analysis of column value and data format description (.txt or .csv) and syntax scripts (.R).
  The external collaborators, especially those involved in validation cohorts, may have access to data upon request.
  With the acceptance of the principal investigator, Rovira i Virgili University's institutional service will guarantee digital access to repositories with raw data generated in research analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once decided the repository web address.
Access Criteria: Decided by the principal investigator.

REFERENCES:
- [Derived] Jimenez-Franco A, Castane H, Martinez-Navidad C, Placed-Gallego C, Hernandez-Aguilera A, Fernandez-Arroyo S, Samarra I, Canela-Capdevila M, Arenas M, Zorzano A, Hernandez-Alvarez MI, Castillo DD, Paris M, Menendez JA, Camps J, Joven J. Metabolic adaptations in severe obesity: Insights from circulating oxylipins before and after weight loss. Clin Nutr. 2024 Jan;43(1):246-258. doi: 10.1016/j.clnu.2023.12.002. Epub 2023 Dec 6. PMID 38101315